CLINICAL TRIAL: NCT05603377
Title: Neuro Anatomical Correlation of Oropharyngeal Swallowing Revisited in Cerebrovascular Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Azhar Elsayed Ali, assistant lecturer of phoniatrics, ENT department Sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-22-10-18
Record Dates: First submitted 2022-10-16; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Other)
  Interventions: Diagnostic Test: functional endoscopic evaluation of swallow

INTERVENTIONS:
Diagnostic Test: functional endoscopic evaluation of swallow — functional endoscopic evaluation of swallow

SUMMARY:
Stroke, main cause of disability in adults, is thought to be the primary cause of swallowing difficulty (dysphagia). Dysphagia is one of the common physical condition among patients with stroke, affecting the large number of stroke patients in the world. It is reported that the occurrence rate of post-stroke dysphagia (PSD) is varies widely, ranging from 19% to 81%, the reason may be associated with the type of stroke, the assessment tools, the timing of the assessment, and so on .Dysphagia is associated with pneumonia, malnutrition, dehydration, increased mortality, and poor long-term outcome. It has been shown that early detection of dysphagia allows for immediate intervention and thereby reduces morbidity, duration of hospitalization, and overall health care costs. Oropharyngeal dysphagia (OD) can have a high impact on the general health of affected patients and can produce two main types of complications in patients with post stroke: (1) those caused by impaired efficacy of swallow, present in 25%-75% of patients, which leads to malnutrition and dehydration and (2) impaired safety of swallow which leads to tracheobronchial aspiration that may cause pneumonia in 50% of cases. Both OD and aspiration are highly prevalent conditions in patients with stroke . Dysphagia is more common in hemorrhagic stroke compared with ischemic stroke, so far, most studies have focused on the latter, presumably due to its higher incidence .The recognition of a brain lesion pattern associated with oropharyngeal dysphagia could help to distinguish those patients in need of more in-depth evaluation and the subsequent adoption of preventive measures. However, it is difficult to predict which patients are susceptible to developing swallowing alterations depending on neuroimaging findings. However, the findings have been inconsistent, mainly due to simplification in the classification of brain injuries into a small number of groups, or to the different methods employed in assessing swallowing function

ELIGIBILITY:
Inclusion Criteria:

- Adult patients> (18 years). Conscious patients Stroke patients confirmed by brain imaging Stroke in the acute and sub-acute phase

Exclusion Criteria:

* Previous stroke Non stroke dysphagia History of other neurologic disorders other than cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
oral phase of swallow | within 7 days
  if there is residue in oral phase of swallow with fluids ,semisolids ,solids
pharyngeal phase of swallow | within 7 days
  if there is residue or penetration or aspiration post swallow with fluids ,semisolids, solids
brain imaging computed tomography CT or magnetic resonance imaging MRI | within 7 days
  brain imaging computed tomography CT or magnetic resonance imaging MRI correlation with oral phase and pharyngeal phase of swallow

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abd-Allah F, Khedr E, Oraby MI, Bedair AS, Georgy SS, Moustafa RR. Stroke burden in Egypt: data from five epidemiological studies. Int J Neurosci. 2018 Aug;128(8):765-771. doi: 10.1080/00207454.2017.1420068. Epub 2018 Jan 4. PMID 29258372
- [Background] Hess F, Foerch C, Keil F, Seiler A, Lapa S. Association of Lesion Pattern and Dysphagia in Acute Intracerebral Hemorrhage. Stroke. 2021 Aug;52(9):2921-2929. doi: 10.1161/STROKEAHA.120.032615. Epub 2021 May 18. PMID 34000833
- [Background] Meng PP, Zhang SC, Han C, Wang Q, Bai GT, Yue SW. The Occurrence Rate of Swallowing Disorders After Stroke Patients in Asia: A PRISMA-Compliant Systematic Review and Meta-Analysis. J Stroke Cerebrovasc Dis. 2020 Oct;29(10):105113. doi: 10.1016/j.jstrokecerebrovasdis.2020.105113. Epub 2020 Jul 9. PMID 32912517
- [Background] Wilmskoetter J, Bonilha L, Martin-Harris B, Elm JJ, Horn J, Bonilha HS. Mapping acute lesion locations to physiological swallow impairments after stroke. Neuroimage Clin. 2019;22:101685. doi: 10.1016/j.nicl.2019.101685. Epub 2019 Jan 22. PMID 30711683